CLINICAL TRIAL: NCT03045315
Title: Are LXRs Involved in Regulation of Human Oocyte Meiosis Resumption?
Brief Title: LXR and Oocyte Meiosis Resumption
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: CHU-303
Record Dates: First submitted 2017-01-27; First posted 2017-02-07 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female

ARMS (1):
- women included in a IVF program (Experimental)
  Interventions: Other: IVF Procedure

INTERVENTIONS:
Other: IVF Procedure

SUMMARY:
Previous studies in animal model showed clearly that lipid homeostasis influence oocyte meiosis resumption. However Liver X Receptors pathway has never been investigated in human ovocyte

DETAILED DESCRIPTION:
In mice deficient of Liver X Receptor (LXR) genes, the oocytes are unable to resume meiosis. Oxysterols are molecules derived from the cholesterol synthesis pathway. They are ligands of the liver X receptors (LXRs). In human, the LXR signalling pathway has never been investigated in this process. The Investigator propose to analyse in granulosa cells surrounding ovocyte the expression of LXR, their target genes and the enzymes involved in oxysterols synthesis. These granulosa cells are normally retrieved and destroyed 18 hours after sperm insemination of oocytes in a In Vitro Fertilization program. The oocyte meiosis resumption will be considered as positive (Granulosa cell positive, GC+) if a zygote is observed 18 hours after sperm insemination and negative (Granulosa cell negative, GC-) if none zygote appears. Moreover the investigator will analyse the quality of embryo development during 5 days after zygote is formed (normal process of In Vitro Fertilization) . The both populations of granulosa cells (GC+ and GC-) will be compared. The measurements of Liver X Receptor genes and the enzymes involved in oxysterols pathways xill be performed by Reverse Transcription-Polymerase Chain Reaction. The accumulation of lipid in granulosa cells will be measures by oil red staining. By this sudy the investigator will probably find new biological markers of resumption meiosis for women enrolled in In Vitro Fertilization programm. Moreover, data will help to better understand the physiopathology of oocyte meiosis failures.

ELIGIBILITY:
Inclusion Criteria:

* woman aged less 37 years
* included in a IVF program
* tubal infertility
* ovarian stimulation with recombinant FSH
* induced ovulation by recombinant chorionic gonaotrophin

Exclusion Criteria:

* dysovulation
* male infertility
* Ovarian insuficiency

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Expression of RNAs of LXR pathways in granulosa cells surrounding oocyte | at day 1
  The day of the retrieve of granulosa cells, RNA extraction will be performed and the expression of Liver X Receptors genes, their downstream target genes and the enzymes of oxyterols synthesis will be analysed.

SECONDARY OUTCOMES:
Accumulation of lipid in granulosa cells surrounding oocyte | at day 5
  Embryo development of inseminated ovocytes at day 5 after sperm insemination during In Vitro Fertilization process

CONTACTS AND LOCATIONS:
Overall Officials: Florence BRUGNON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France